CLINICAL TRIAL: NCT00360789
Title: The Effects of Standardized Physical Therapy and Functional Strength Training on Upper Limb Function and Neuromuscular Weakness After Stroke: a Pilot Study
Brief Title: Evaluation of Whether Functional Strength Training Can Enhance Motor Recovery of the Upper Limb After Stroke
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St George's, University of London (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GR070116MA
Record Dates: First submitted 2006-08-03; First posted 2006-08-07 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2006-08

CONDITIONS: Stroke
Keywords: STROKE REHABILITATION; pHYSICAL THERAPY
MeSH Terms: conditions — Stroke

INTERVENTIONS:
Behavioral: Conventional UK physical therapy
Behavioral: Increased intensity of UK conventional physical therapy (PT)
Behavioral: UK conventional PT plus functional strength training

SUMMARY:
The purpose of this study is to test the hypothesis that adding functional strength training to UK conventional therapy improves muscle function and walking than either UK conventional therapy alone or increased intensity of UK conventional therapy.

DETAILED DESCRIPTION:
Neuromuscular weakness occurs frequently after stroke and the processes underlying recovery are still poorly understood. Accepted practice in UK physiotherapy is to avoid training of muscle strength after stroke but there is preliminary evidence that it might be effective.

An observer-blind randomised pilot clinical trial (Phase II). Subjects will be within 3 months of first stroke with some voluntary movement in the paretic upper limb.

A Research Physiotherapist, blinded to measurement, will recruit subjects, allocate subjects to one of three intervention groups using sequentially numbered sealed envelopes containing previously allocated intervention cards and provide interventions. Ten participants will be recruited to each group therefore the trial will recuit 30 participants. The Research Assessor, blinded to intervention allocation will undertake all measurements.

Conventional therapy (control) will be provided as normal for the clinical setting, the additional conventional therapy (experimental 1)or functional strength training (experimental 2) will be provided for one hour, five times a week for six weeks. Subjects in the two experimental groups will also receive the conventional therapy standard in their clinical setting.

Blinded measurement will be made before randomisation, at the end of intervention and 12-weeks thereafter. Primary outcomes are the Action Research Arm Test (ARAT)and the Nine Hole Peg Test (9HPT). The secondary outcomes are peak torque around the elbow joint in elbow flexion and extension, grip force, pinch force, smoothness of movement during turning a cranked wheel and reciprocal inniveration of biceps and triceps during turning of a cranked wheel.

Data will be analysed using descriptive statistics and the estimation of standard deviations will be used to inform a power calculation to estimate sample size for a Phase II randomised controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Be between one week and three months after stroke when recruited to the study
* Have some voluntary muscle activity in the paretic upper limb

Exclusion Criteria:

* Obvious unilateral visuospatial neglect
* Upper limb movement deficits attributable to non-stroke pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-06; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Action Research Arm Test (ARAT)
Nine Hole Peg Test (9HPT)

SECONDARY OUTCOMES:
peak torque around the elbow joint in elbow flexion and extension
grip force
pinch force
smoothness of movement during turning a cranked wheel
reciprocal inneveration of biceps and triceps during turning of a cranked wheel.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie M Pomeroy, PhD, Study Chair — St George's, University of London
Locations (1):
- St George's Hospital NHS Trust, London, United Kingdom